CLINICAL TRIAL: NCT02310451
Title: Pilot Study of Exosomes Before and After BRAF Inhibitor Therapy in Patients With Advanced Unresectable or Metastatic BRAF Mutation-positive Melanoma
Brief Title: Study of Molecular Mechanisms Implicated in the Pathogenesis of Melanoma. Role of Exosomes
Acronym: EXOSOMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-AOI-10
Record Dates: First submitted 2014-11-13; First posted 2014-12-08 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metastatic melanoma (Experimental): Patients affected by advanced melanoma not resectable (stage IIIc) or metastatic (stage IV)
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — blood test to J0-M3-M6-M12

SUMMARY:
Recent progresses have been made in the treatment of metastatic melanoma, nevertheless improved patient survival is still limited because of primary resistance and relapses. It is therefore important to continue to understand the molecular mechanisms involved in melanoma development and progression to improve the management of patients.

Drugs such as the alkylating agents (temozolomide and fotemustine) or vemurafenib trigger senescence-like phenotypes in melanoma cells. It is now known that senescent cells secrete some factors that exert a pro-tumoral role but the potential existence and the role of insoluble factors remain undetermined.

Preliminary results from the investigators laboratory indicate the presence in the senescent secretome of exosomes; microvesicles involved in intercellular communication, immunomodulatory functions, and tumorigenesis. Several studies showed that these vesicles shape the tumor microenvironment and contribute to the migration of cancer cells.

Their interest in oncology as a prognostic factor and marker of therapeutic response is increasing.

Thus, our project aims to study the effect of exosomes produced by senescent melanoma cells in the development and progression of melanoma in vitro and in vivo using cell cultures and animal models.

In addition, the investigator propose a pilot study whose objective is to determine the effect of vemurafenib on nanovesicles produced by patients with advanced unresectable or metastatic melanoma.

The investigator hope to show that exosomes participate in the process of drug resistance and relapse, with the goal of developing (with the exosomes study) theranostic tools for personalized care in patients.

DETAILED DESCRIPTION:
Metastatic melanoma is an aggressive tumor with a 5-year survival rate of about 6 months. Although recent progresses have been made in the treatment of metastatic melanoma, improved patient survival is still limited because of primary resistance and relapses. It is therefore important to continue to understand the molecular mechanisms involved in melanoma development and progression to improve current treatments and / or to discover new anti-metastatic melanoma treatments.

Drugs such as the alkylating agents (temozolomide and fotemustine) or vemurafenib trigger senescence-like phenotypes in melanoma cells. Although senescence is a process that limits the proliferation of cells, it is now known that senescent cells secrete factors that exert a pro-tumoral role. If many studies have focused on the role of the soluble factors of this secretome, the potential existence and the role of insoluble factors remain undetermined. Preliminary results from the investigators laboratory indicate the presence in the senescent secretome of exosomes; microvesicles involved in intercellular communication, immunomodulatory functions, and tumorigenesis. The exovesicules discharged by a cell in its environment are the subject of increasing interest in oncology as a prognostic factor and marker of therapeutic response. Several studies showed that these vesicles shape the tumor microenvironment and contribute to the migration of cancer cells.

This project aims to study the effect of exosomes produced by senescent melanoma cells in the development and progression of melanoma in vitro and in vivo using cell cultures and animal models. In addition, the investigator propose a pilot study whose objective is to determine the effect of vemurafenib on production, quantity, size and composition of nanovesicles produced by patients with advanced unresectable or metastatic melanoma. The investigator hope to show that exosomes participate in the process of drug resistance and relapse, with the goal of developing (with the exosomes study) theranostic tools for personalized care in patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sexes at least 18 years of age
* Patient with advanced melanoma unresectable (stage IIIc) or metastatic (stage IV)
* Patient for whom is considered a systemic treatment by BRAF inhibitor
* Patient no previously treated or no responding to chemotherapy with a last injection> 1month
* Patient affected by a melanoma measurable according to version 1.1 of RECIST criteria
* Patient with a life expectancy superior than 3 months
* Serum pregnancy test negative for all women of childbearing age
* ECOG ≤1
* Patient affiliated to French social security
* Patient able to understand and communicate with the investigator and to comply with the requirements of the study
* Patient must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations

Exclusion Criteria:

* Patients not eligible to a BRAF inhibitor therapy or affected by a serious disease wich could require a treatment susceptible to interfere with melanoma treatment
* Pregnant and lactating women
* Patient with active malignancy or a previous malignancy within the past 3 years; except for patient with resected BCC, resected cutaneous SCC, resected carcinoma in-situ of the cervix, and resected carcinoma in-situ of the breast
* Past medical history record of infection with human immunodeficiency virus or viral hepatite C or B
* Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
number of exosomes | change from Day 0 at Month12
  Measure of the number of exosomes (µg of proteins or particles)/ml in peripheral blood by differential ultracentrifugation before and after treatment.

SECONDARY OUTCOMES:
number of patient with a detection test of exosomes positive measured | change from Day 0 at Month12
  Calculation of number of patients with a detection test of exosomes positive measured in the peripheral blood after differential ultracentrifugation by protein assay and Nanosight before and after treatment.
survival | Month 12
  Difference in survival (overall survival and progression frre-survival) between patients depending on the size and number of exosomes (µg of proteins or particles)/ml before and after treatment, according to the method of Kaplan Meier
Tumoral response | Month 12
  Difference of tumoral response (RECIST criteria) between patients depending on variation of the number of exosomes (µg of proteins or particles)/ml, size and composition before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henri MONTAUDIE, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice ^Hôpital de l'Archet, Nice, France